CLINICAL TRIAL: NCT02635269
Title: Fat and Sugar Metabolism During Exercise in Patients With Metabolic Myopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Karen Lindhardt Madsen, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Metabolic Myopathy; H-15015150 (Other: De Videnskabsetiske Komiteer for Region Hovedstaden)
Record Dates: First submitted 2015-12-09; First posted 2015-12-18 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Metabolism, Inborn Errors; Lipid Metabolism, Inborn Errors; Carbohydrate Metabolism, Inborn Errors; Long-Chain 3-Hydroxyacyl-CoA Dehydrogenase Deficiency; Glycogenin-1 Deficiency (Glycogen Storage Disease Type XV); Carnitine Palmitoyl Transferase 2 Deficiency; VLCAD Deficiency; Medium-chain Acyl-CoA Dehydrogenase Deficiency; Multiple Acyl-CoA Dehydrogenase Deficiency; Carnitine Transporter Deficiency; Neutral Lipid Storage Disease; Glycogen Storage Disease Type II; Glycogen Storage Disease Type III; Glycogen Storage Disease Type IV; Glycogen Storage Disease Type V; Muscle Phosphofructokinase Deficiency; Phosphoglucomutase 1 Deficiency; Phosphoglycerate Mutase Deficiency; Phosphoglycerate Kinase Deficiency; Phosphorylase Kinase Deficiency; Beta Enolase Deficiency; Lactate Dehydrogenase Deficiency; Glycogen Synthase Deficiency
Keywords: Ergometry; Stable isotope tracers
MeSH Terms: conditions — Metabolism, Inborn Errors; Lipid Metabolism, Inborn Errors; Carbohydrate Metabolism, Inborn Errors; Trifunctional Protein Deficiency With Myopathy And Neuropathy; Carnitine palmitoyl transferase 2 deficiency; VLCAD deficiency; Medium chain acyl CoA dehydrogenase deficiency; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Systemic carnitine deficiency; Chanarin-Dorfman Syndrome; Glycogen Storage Disease Type II; Glycogen Storage Disease Type III; Glycogen Storage Disease Type IV; Glycogen Storage Disease Type V; Glycogen Storage Disease Type VII; Glycogen Storage Disease XIV; Dimauro disease; Phosphoglycerate Kinase 1 Deficiency; Glycogen Storage Disease Type Ix; Glycogen Storage Disease XIII; Lactate Dehydrogenase Deficiency | interventions — Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sugar (Experimental): The subjects exercise on the cycle-ergometer until exhaustion or for a maximum of 1 hour at an intensity that corresponds to 60-65% of VO2max.
  Interventions: Other: Sugar

INTERVENTIONS:
Other: Sugar — 10 minutes before exercising, the subjects are given a bolus of glucose solution 0.2 g/kg in a cubital vein catheter and a constant infusion of 10% glucose solution is started (100ml/h). The infusion continues throughout the exercise period.
  Other Names: 10 % glucose infusion

SUMMARY:
This study aims to characterize the pathophysiological mechanisms of 21 different metabolic myopathies. The study will focus on exercise capacity and the metabolic derangement during exercise.

DETAILED DESCRIPTION:
Patients will be compared to a group of matched healthy control subjects (matched for age, gender, physical activity level and BMI) for comparison of the primary and secondary outcome measures.

Methods:

Each subject will go through 3 test days.

Test day 1:

* International Physical Activity Questionnaire (IPAQ). The results will be used to match the patients to control subjects.
* DEXA-scan. This is used to estimate the volume of distribution for stable isotope tracers.
* Maximal oxidative capacity test (max-test). On a cycle ergometer, subjects will exercise for approximately 15 minutes with increasing resistance until exhaustion. The peak oxidative and workload capacities will be compared to the healthy controls and will be used to find the workload that corresponds to 55-65 % of VO2max used in the following exercise tests.
* Blood samples. Samples will be drawn before exercise and at exhaustion and will be analyzed for the plasma concentrations of glucose, lactate, ammonia, creatine kinase and myoglobin.

Test day 2:

•Long exercise test #1. The purpose of this test is to measure the total fat and sugar oxidation rates during exercise by using stable isotope tracers.

Subjects arrive at the laboratory after 3-9 hours of fasting. One IV-catheter is inserted in the cubital vein in one arm and another in a peripheral vein in the other hand. The stable isotope tracers will be given in the cubital vein as a constant infusion of solutions of:

* [U-13C]-palmitate (0.0026 mg x kg-1 x min-1, after a priming bolus of 0.085 mg x kg-1 NaH13CO3)
* [1,1,2,3,3-2H5]-glycerol (0.0049 mg x kg-1 x min-1 )
* [6.6-2H2]-glucose (0.0728 mg x kg-1 x min-1 ) For two hours the subjects rests while receiving the infusions until the tracers have distributed in the body and reached a steady state. After the rest, the subjects exercise on the cycle-ergometer until exhaustion or for a maximum of 1 hour at an intensity that corresponds to 55-65% of VO2max.

The heart rate is continuously measured during exercise, and every other minute the subject evaluates his/her degree of exertion (Rate of Perceived Exertion, RPE) on a Borg scale.

•Blood and breath samples From 20 minutes before exercise and every ten minutes until the end of exercise, blood samples are drawn and samples of the expired breath are collected.The breath is analysed for 13CO2 -enrichment. The blood is analysed for the plasma concentrations of glucose, lactate, ammonia, creatine kinase and myoglobin.

Test day 3:

•Long exercise test #2. The purpose of this test is to investigate exercise capacity and performance measured as HR, VO2 and RPE during prolonged exercise. To mimic the conditions for the working muscles in healthy persons who have an intact metabolism, the patients are given an infusion of a 10% glucose solution to maintain the blood sugar while exercising.

Subjects arrive at the laboratory after 3-9 hours fasting. After 2 hours of rest, the subjects exercise on the cycle-ergometer until exhaustion or for a maximum of 1 hour at an intensity that corresponds to 60-65% of VO2max, like they did on test day 2. This time the subjects are not given stable isotope tracers. 10 minutes before exercising, the subjects are given a bolus of glucose solution 0.2 g/kg in a cubital vein catheter and a constant infusion of 10% glucose solution is started (100ml/h). The infusion continues throughout the exercise period.

Assessments of heart rate, Rate of Perceived Exertion and blood sampling follow the same protocol as on test day 1, except no breath samples are taken and no analyses of stable isotopes are made, since the tracers are not used on test day 3.

* Blood samples. From 20 minutes before exercise and every ten minutes until the end of exercise, blood samples are drawn. The blood is analysed for the plasma concentrations of glucose, lactate, ammonia, creatine kinase and myoglobin.
* Muscle Biopsy At the end of test day 1 the investigators will perform a voluntary muscle biopsy.

Statistical Methods:

The investigators will use a paired t-test, two-tailed testing (or the corresponding non-parametric test, if the assumption of normality is not met). A p-value of < 0.05 will be considered significant. Results will be reported with Confidence Intervals of the difference in means. SigmaPlot version 11.0 (or a similar statistical program) will be used for statistical analysis.

No interim analyses will be made during the 4 days trial period. In the case, that a patient withdraws/is withdrawn, the obtained data from the completed tests will be included in the analyses. Raw data that is clearly and indisputably a result of an error in measurement will not be included (evaluated by the investigator). Missing or lost data will if possible be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with genetically and/or biochemically verified LCHAD Deficiency
* Healthy controls needs to be healthy to be included, evaluated by the investigator.

Exclusion Criteria:

* Competing conditions at risk of compromising the results of the study.
* Pregnancy or breastfeeding
* Cardiac or pulmonary disease contraindicating peak exercise testing or strenuous exercise.
* Inability to understand the purpose of the trial or corporate for the conduction of the experiments.
* Veins that are too difficult to puncture for blood sampling or insertion of intravenous catheters, evaluated by the investigator
* Moderate to severe muscle weakness, that prevents the subject completing 10 minutes of cycle-ergometry exercise at 60-70 % of VO2peak, evaluated by the investigator.
* Participation in other trials that may interfere with the results.
* Intake of medications that may interfere with the results or may compromise exercise performance, as evaluated by the investigators.
* Donation of blood within 30 days prior to conduction of the tests on test day 1.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Total fat oxidation (rate of disappearance) during prolonged moderate intensity exercise. Measured as micro mol per kg per minute. | Measured at at time (minutes) -120, -20, -10, 0, 10, 20, 30, 40, 50, 60. Zero is the indicatet start of 1 hour cycling test. Measured on day 2 of participation
  Measured using stable isotope technique ([U-13C]-palmitate, [1,1,2,3,3-2H5]-glycerol and [6.6-2H2]-glucose ) and indirect calorimetry.

SECONDARY OUTCOMES:
Maximal oxidative capacity (mL*kg-1*minutes-1) | Day 1 of participation
  Oxidative capacity is measured continuously during a maximum exercise test on the first day of the trial. The test lasts about 15 minutes (when the participant is fully exhausted). The maximal oxidative capacity is the peak measure during the test.
Endurance measured as minutes:seconds | Day 2 and 4 of participation
  During 1 hour cycling test 1 and 1 hour cycling test 2 on day 2 and 4 of participation. The test will last for 1 hour or until exhaustion. Endurance will be defined as the total exercise duration.
Heart rate (HR) during prolonged exercise, with and without blood sugar maintained by an infusion of a 10% glucose solution. Measured in beats per minute. | During 1 hour cycling test 1 and 1 hour cycling test 2 on day 2 and 4 of participation.
  During 1 hour cycling at 55-65% of VO2max the heart rate is measured every 2 minuts.
Oxygen consumption rate (VO2) during prolonged exercise, with and without blood sugar maintained by an infusion of a 10% glucose solution. Measured in mL. | During 1 hour cycling test 1 and 1 hour cycling test 2 on day 2 and 4 of participation.
  During 1 hour cycling at 55-65% of VO2max the oxygen consumption rate is continuously measured.
Self-evaluated exertion (Rate of Perceived Exertion (RPE)) during prolonged exercise, with and without blood sugar maintained by an infusion of a 10% glucose solution. Measured using a Borg-scale (6-20). | During 1 hour cycling test 1 and 1 hour cycling test 2 on day 2 and 4 of participation.
  During 1 hour cycling at 55-65% of VO2max the participant is asked to rate their exertion every 2 minutes.
Maximal workload capacity. Measured in watt | Day 1 of participation
  The participant will be cycling at incremental workload until exhaustion. The test lasts about 15 minutes (when the participant is fully exhausted). The maximal workload is the peak measure at the end of the test.
Total glucose oxidation (rate of disappearance) during prolonged moderate intensity exercise. Measured as micro mol per kg per minute. | Measured at at time (minutes) -120, -20, -10, 0, 10, 20, 30, 40, 50, 60. Zero is the indicatet start of 1 hour cycling test. Measured on day 2 of participation
  Measured using stable isotope technique ([U-13C]-palmitate, [1,1,2,3,3-2H5]-glycerol and [6.6-2H2]-glucose ) and indirect calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Madsen, MD, Principal Investigator — Neuromuscular Research Unit
Locations (1):
- Neuromuscular Research Unit, 3342, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oldfors A, DiMauro S. New insights in the field of muscle glycogenoses. Curr Opin Neurol. 2013 Oct;26(5):544-53. doi: 10.1097/WCO.0b013e328364dbdc. PMID 23995275
- [Background] Liang WC, Nishino I. State of the art in muscle lipid diseases. Acta Myol. 2010 Oct;29(2):351-6. PMID 21314018
- [Background] Orngreen MC, Duno M, Ejstrup R, Christensen E, Schwartz M, Sacchetti M, Vissing J. Fuel utilization in subjects with carnitine palmitoyltransferase 2 gene mutations. Ann Neurol. 2005 Jan;57(1):60-6. doi: 10.1002/ana.20320. PMID 15622536
- [Derived] Raaschou-Pedersen D, Madsen KL, Stemmerik MG, Eisum AV, Straub V, Vissing J. Fat oxidation is impaired during exercise in lipin-1 deficiency. Neurology. 2019 Oct 8;93(15):e1433-e1438. doi: 10.1212/WNL.0000000000008240. Epub 2019 Sep 6. PMID 31492716
- [Derived] Madsen KL, Stemmerik MG, Buch AE, Poulsen NS, Lund AM, Vissing J. Impaired Fat Oxidation During Exercise in Long-Chain Acyl-CoA Dehydrogenase Deficiency Patients and Effect of IV-Glucose. J Clin Endocrinol Metab. 2019 Sep 1;104(9):3610-3613. doi: 10.1210/jc.2019-00453. PMID 30990523